CLINICAL TRIAL: NCT01432795
Title: Gliding Aids for Medical Compression Stockings - Practicability in Elderly Patients With Chronic Venous Insufficiency
Brief Title: Practicability of Gliding Aids for Medical Compression Stockings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: JH Rahn Foundation, Zurich (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH2010-0329/5
Record Dates: First submitted 2011-05-02; First posted 2011-09-13 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Venous Insufficiency; Post-thrombotic Syndrome
Keywords: chronic venous insufficiency; post-thrombotic syndrome; medical compression therapy; compression stocking; gliding aid; stocking butler; adherence to treatment
MeSH Terms: conditions — Postthrombotic Syndrome; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test series of 6 types of gliding aids (Experimental): Each study subjects tests a series of gliding aids or stocking butlers:
  * 4 gliding aids
  * 2 stocking "butlers", one with and without handle
  * 3 medical compression stockings with open tip, compression class 3 (36-46mmHg)
  * 3 medical compression stockings w. closed tip, compression class 3 (36-46mmHg)
  * 2 superimposed stockings with closed tip, compression class 1 (18-21 mmHg)
  Interventions: Device: Gliding aids for medical compression stockings

INTERVENTIONS:
Device: Gliding aids for medical compression stockings — Each subject tests devices:
  * 3 gliding aids for stockings with closed tips
  * 3 gliding aids for stockings with open tips
  * 2 stocking butlers using
  * 3 medical compression stockings with open tip, compression class 3 (36-46mmHg)
  * 3 medical compression stockings w. closed tip, compression class 3 (36-46mmHg)
  * 2 superimposed compression stockings class 1 (18 - 21 mmHg)
  Other Names: Gliding aids:; Easy Slide (Sigvaris); Easy Slide Caran (Sigvaris); Venotrain Glider (Bauerfeind); Blue Standard Foot Slip (Bauerfeind); Easy Glide (Eureka) (Salzmann); Socks Jet with and without handle (Salzmann); Mediven Butler (Cosanum)

SUMMARY:
Medical compression stockings are highly effective in the prevention, treatment, and secondary prevention of chronic venous insufficiency and of post-thrombotic syndrome. Non-adherence to the prescribed compression treatment concerns approximately 40% of patients. Elderly patients are often unable to handle stockings in order to put them on properly in the morning and to undress in the evening. Gliding aids and stocking "butlers" are two types of tools to facilitate the dressing manoeuvre with medical stockings.

The present study evaluates four different gliding aids and two different stocking "butlers" to put on three different types of compression stockings. The study is conducted with forty consenting subjects with advanced chronic venous insufficiency.

DETAILED DESCRIPTION:
Subjects: 40 consenting patients >65y old, with CEAP C4-6 chronic venous insufficiency

Stockings:

One class 3 (36 - 46 mmHg interface pressure) with closed tip One class 3 with open tip Two superimposed class 1 (18 - 21 mmHg)

Gliding aids and stocking "butlers" Three types of gliding aids for closed tip stockings Three types of gliding aids for open tip stockings Two types of stocking "butlers", one optional with mounted handles

ELIGIBILITY:
Inclusion Criteria:

> 65 years old Chronic venous insufficiency CEAP C4-6

Exclusion Criteria:

Dementia Blindness Paraplegia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of successfully dressed medical stockings per subject | Per subject: 120 minutes (one "run"); to complete the whole study (40 subjects): 14 months
  The primary end point is straight: The medical stocking is dressed (at the patient's leg) or it is not dressed. Each gliding aid and each stocking "butler" is tested with this end point.

SECONDARY OUTCOMES:
Patient satisfaction by gliding aid or stocking butler (score) | Per subject 120 minutes (one "run"); to complete the whole study (40 subjects): 14 months
  Patients are asked to score each gliding aid and each stocking "butler" with a mark between "1" (bad) and "6" (very good).

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Hafner, Professor, Principal Investigator — Department of Dermatology, University Hospital of Zurich, Switzerland
Locations (1):
- Department of Dermatology, University Hospital of Zurich, Switzerland, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Sippel K, Seifert B, Hafner J. Donning devices (foot slips and frames) enable elderly people with severe chronic venous insufficiency to put on compression stockings. Eur J Vasc Endovasc Surg. 2015 Feb;49(2):221-9. doi: 10.1016/j.ejvs.2014.11.005. Epub 2015 Jan 8. PMID 25579875